CLINICAL TRIAL: NCT00506389
Title: A Six-Week Double-Blind Randomized, Placebo-Controlled, Parallel Group, Efficacy and Safety, Sleep Lab Trial With Org 50081 in Patients With Chronic Primary Insomnia
Brief Title: A Six Week, Double-Blind Randomized, Efficacy and Safety, Sleep Lab Trial With Esmirtazapine (Org 50081) (P05707)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05707; 176002 (Other: Organon)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Insomnia
Keywords: Sleep Initiation and Maintenance Disorders, Sleep Disorders, Intrinsic Dyssomnias, Sleep Disorders, Nervous System Diseases, Mental Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Nervous System Diseases; Mental Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esmirtazapine 3.0 mg (Experimental): Participants took placebo tablets on Days -7 and -6, esmirtazapine 3.0 mg tablets on Days 1-42, and placebo tablets on Days 43-50. Tablets were taken by mouth once daily in the evening.
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 4.5 mg (Experimental): Participants took placebo tablets on Days -7 and -6, esmirtazapine 4.5 mg tablets on Days 1-42, and placebo tablets on Days 43-50. Tablets were taken by mouth once daily in the evening.
  Interventions: Drug: Esmirtazapine
- Placebo (Placebo Comparator): Participants took placebo tablets on Days -7 and -6, placebo tablets on Days 1-42, and placebo tablets on Days 43-50. Tablets were taken by mouth once daily in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmirtazapine — Esmirtazapine maleate was provided as tablets for oral use containing 3.0 mg, or 4.5 mg of active compound. In addition, tablets contain the following excipients: hydroxypropyl cellulose, maize starch (United States Pharmacopeia [USP] name corn starch), magnesium stearate, and lactose monohydrate.
  Other Names: ORG 50081
  Arms: Esmirtazapine 3.0 mg; Esmirtazapine 4.5 mg
Drug: Placebo — The placebo tablets contained the following excipients: hydroxypropyl cellulose, maize starch (USP name corn starch), magnesium stearate, and lactose monohydrate.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the efficacy, safety and tolerability of esmirtazapine (Org 50081) compared to placebo in patients with chronic primary insomnia.

DETAILED DESCRIPTION:
Insomnia is a common complaint or disorder throughout the world. About one third of the population in the industrial countries reports difficulty initiating or maintaining sleep, resulting in a non-refreshing or non-restorative sleep. The majority of the insomniacs suffer chronically from their complaints. It has been reported that in patients with chronic insomnia lasting longer than six months, 50% had a past or current mental disorder. This raises the possibility that treatment of insomnia may reduce the risk for psychological conditions. This double-blind, placebo-controlled, parallel, randomized clinical trial is designed to assess the efficacy and safety of esmirtazapine in patients suffering from chronic primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of chronic primary insomnia

Exclusion Criteria:

* Other sleep disorder such as sleep apnea, restless leg syndrome, narcolepsy, sleep/wake rhythm disorders
* Has significant medical or psychiatric illness as causing the sleep disorder
* Diagnosed with major depressive disorder
* Substance abuse within the past year
* Night worker or work on rotating shifts
* Has had serious head injury, stroke, epilepsy
* Has a history of bipolar disorder or family (immediate family) history of suicide
* Smokes more than 15 cigarettes per day and cannot abstain from smoking during the night or in the sleep laboratory
* Drinks beverages containing more than 500 mg caffeine per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2007-06-06 (Actual); Primary Completion 2008-02-13 (Actual); Study Completion 2008-02-13 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ivgy-May N, Ruwe F, Krystal A, Roth T. Esmirtazapine in non-elderly adult patients with primary insomnia: efficacy and safety from a randomized, 6-week sleep laboratory trial. Sleep Med. 2015 Jul;16(7):838-44. doi: 10.1016/j.sleep.2015.04.001. Epub 2015 Apr 16. PMID 26047892

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmirtazapine 3.0 mg: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, esmirtazapine 3.0 mg tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. After this, participants were followed for safety up to Day 50 during the Follow-Up Period.
- Esmirtazapine 4.5 mg: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, esmirtazapine 4.5 mg tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. After this, participants were followed for safety up to Day 50 during the Follow-Up Period.
- Placebo: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, placebo tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. After this, participants were followed for safety up to Day 50 during the Follow-Up Period.
Period: In-treatment Period
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Started | 143 | 139 | 137
All Participants Treated | 139 | 138 | 136
Completed | 117 | 124 | 125
Not Completed | 26 | 15 | 12
Not completed — Other | 3 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Lack of compliance | 1 | 0 | 0
Not completed — Reasons not related to trial | 4 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 4
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Adverse Event | 11 | 5 | 2
Not completed — Randomized but not treated | 4 | 1 | 1
Period: Follow-up Period
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Started | 139 (22 participants who discontinued treatment entered the Follow-up Period.) | 138 (14 participants who discontinued treatment entered the Follow-up Period.) | 136 (11 participants who discontinued treatment entered the Follow-up Period.)
Completed | 139 | 138 | 136
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo | Total
Number analyzed (Participants) | 143 | 139 | 137 | 419
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (11.3) | 44.5 (11.5) | 46.6 (10.5) | 44.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 89 | 90 | 277
  Male | 45 | 50 | 47 | 142

OUTCOME MEASURES:

1. Primary Outcome: Average Wake Time After Sleep Onset (WASO) During the In-Treatment Period
Description: WASO was defined as the total objective time awake after the onset of persistent sleep until the end of the 8-hour sleep cycle period as measured by polysomnography (PSG). WASO was calculated as the mean of Nights 1, 15, and 36.
Time Frame: From Day 1 to Day 36
Population: The Intent-to-Treat (ITT) group consisted of all participants who were randomized, received at least one dose of double-blind trial medication, and had at least one post-randomization efficacy assessment. Fifteen participants from 1 site were excluded from all efficacy analyses.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 133 | 133 | 132
Minutes | 45.6 (25.7) | 45.5 (26.5) | 76.1 (46.0)

2. Secondary Outcome: Average Latency to Persistent Sleep (LPS) During the In-Treatment Period
Description: LPS was defined as the time in minutes from lights out to the first 20 consecutive epochs scored as sleep as measured by PSG. LPS was calculated as the mean of Nights 1, 15, and 36.
Time Frame: From Day 1 to Day 36
Population: The ITT group consisted of all participants who were randomized, received at least one dose of double-blind trial medication, and had at least one post-randomization efficacy assessment. Fifteen participants from 1 site were excluded from all efficacy analyses.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 133 | 133 | 132
Minutes | 28.7 (28.4) | 26.1 (23.0) | 40.5 (27.3)

3. Secondary Outcome: Average Subjective Total Sleep Time (TST) During the In-Treatment Period
Description: TST was defined as the total amount of time in minutes that was actually spent sleeping the previous night as recorded daily in the participant's sleep diary. TST values over the 6 week In-Treatment Period were averaged for each participant, and average TST was then reported by treatment arm. For participants with missing data, the average of the nights for which TST data were available was used in the analysis.
Time Frame: From Day 1 to Day 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 133 | 133 | 132
Minutes | 384.6 (63.6) | 384.6 (66.2) | 351.6 (57.2)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 50
Description: Adverse events (AEs) were monitored for All Participants Treated (receiving at least one dose of study drug) during the 6-week In-treatment Period and the subsequent 1-week Follow-up Period. Six participants did not receive study drug and were not included.
Groups:
- Esmirtazapine 3.0 mg In-treatment: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, esmirtazapine 3.0 mg tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. Tablets were taken by mouth once daily in the evening.
- Esmirtazapine 4.5 mg In-treatment: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, esmirtazapine 4.5 mg tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. Tablets were taken by mouth once daily in the evening.
- Placebo In-treatment: Participants took placebo tablets during the 10- to 14-day Placebo Washout Period, placebo tablets during the 6-week In-treatment Period, and placebo tablets during the 1-week Placebo Withdrawal Period. Tablets were taken by mouth once daily in the evening.
- Esmirtazapine 3.0 mg Follow-up: After participants received placebo tablets during the Placebo Washout Period and 3.0 mg esmirtazapine during the In-treatment Period, participants were followed for safety up to Day 50 during the Follow-up Period.
- Esmirtazapine 4.5 mg Follow-up: After participants received placebo tablets during the Placebo Washout Period and 4.5 mg esmirtazapine during the In-treatment Period, participants were followed for safety up to Day 50 during the Follow-up Period.
- Placebo Follow-up: After participants received placebo tablets during the Placebo Washout Period and placebo during the In-treatment Period, participants were followed for safety up to Day 50 during the Follow-up Period.
Arm/Group | Esmirtazapine 3.0 mg In-treatment | Esmirtazapine 4.5 mg In-treatment | Placebo In-treatment | Esmirtazapine 3.0 mg Follow-up | Esmirtazapine 4.5 mg Follow-up | Placebo Follow-up
Serious Adverse Events (participants affected / at risk) | 0/139 | 1/138 | 0/136 | 0/139 | 0/138 | 0/136
Other Adverse Events (participants affected / at risk) | 20/139 | 24/138 | 13/136 | 2/139 | 1/138 | 1/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 3.0 mg In-treatment (N=139) | Esmirtazapine 4.5 mg In-treatment (N=138) | Placebo In-treatment (N=136) | Esmirtazapine 3.0 mg Follow-up (N=139) | Esmirtazapine 4.5 mg Follow-up (N=138) | Placebo Follow-up (N=136)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 3.0 mg In-treatment (N=139) | Esmirtazapine 4.5 mg In-treatment (N=138) | Placebo In-treatment (N=136) | Esmirtazapine 3.0 mg Follow-up (N=139) | Esmirtazapine 4.5 mg Follow-up (N=138) | Placebo Follow-up (N=136)
Headache (Nervous system disorders) | 5 (7) | 7 (9) | 9 (11) | 2 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 16 (18) | 18 (20) | 4 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the Sponsor, at least 6 weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.